CLINICAL TRIAL: NCT06246188
Title: Use of Stress-CMR Using Regadenoson and GE-267 in Adult Patients with Known or Suspected Coronary Artery Disease Using Mobile Cardiac MRI Units in a Single-arm Open-label Study
Brief Title: Use of Stress-CMR Using Regadenoson and GE-267 in Adult Patients with Known or Suspected Coronary Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: German Heart Institute (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Sebastian Kelle, Univ.-Prof. Dr. med., German Heart Institute
Other Study IDs: RAPS-22-02
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac MRI; Stress perfusion cardiac MRI; Regadenoson; GE-267; Diagnosis; Rural Region; mycocardial perfusion defect; mobile MRI; CMR; Cardiac Magnetic Resonance
MeSH Terms: conditions — Coronary Artery Disease; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Cardiac MRI using Regadenoson and GE-267 — Performing stress-cardiac MRI for clinical diagnostic in adult patients with suspected coronary artery disease

SUMMARY:
Stress cardiac MRI is crucial for diagnosing coronary artery disease in adults. Currently, it is mainly performed with vasodilators in specialized centers. Introducing mobile CMR units could increase accessibility, especially in rural areas, potentially reducing unnecessary invasive procedures. The objectives include demonstrating the feasibility of mobile stress perfusion CMR, detecting CAD using Regadenoson, and evaluating the image quality of GE-267 in real-world scenarios.

DETAILED DESCRIPTION:
Stress-cardiac MRI (CMR) has a Class I indication for the clinical diagnostic workup in adult patients with suspected coronary artery disease (CAD), including those with epicardial as well as microvascular disease (Gulati M et al. 2021; Zeppenfeld et al. 2022). According to large registry data, in more than 90% of stress-CMR-exams the test was performed using a vasodilator (Adenosine/Regadenoson) at tertiary care centers. However, the use of mobile CMR-units would make this high-end diagnostic tool available to much more patients, especially in rural areas, and by this potentially decrease the rate of unnecessary invasive procedures to rule out CAD. Therefore, we define following objectives:

1. Demonstrate the easy performance of stress Perfusion CMR in a mobile setting using a short and patient/user friendly CMR-protocol. Our hypothesis is that there are no differences in performing stress CMR using a mobile setting versus a stationary setting (based on published literature).
2. Detect mycocardial perfusion defect indicating significant CAD using Regadenoson
3. Evaluate the image quality of GE-267 in a real-world setting using a quantitative score-systeme

ELIGIBILITY:
Inclusion Criteria:

Adults with known or suspected coronary artery disease based one of the following criteria:

1. Abnormal CMR without stress in a previous CMR measurement (e.g. new onset of wall motion abnormalities or reduced LVEF)
2. Referral from local cardiologist based on one of the following criteria:

   1. Patients has a diagnosed coronary artery disease based on other methods
   2. Patients has a high-risk profile based on risk stratification using clinical evaluation (ESC-Score > 5%), the assessment of LV function by resting echocardiography, and, in the majority of cases, non-invasive assessment of ischaemia or coronary anatomy.
   3. Patients demonstrate chronic kidney disease (CKD III or higher) and diabetes
   4. Patients demonstrate history of peripheral artery disease (PTA/Stent) or TEA of the carotids or previous operation of atherosclerotic aortic aneurysms

      * Male or female subjects aged ≥18 years
      * Patient fully responsible and can understand/sign the study from a legal aspect

Exclusion Criteria:

* Patient refusal to participate
* Any contraindication to perform an MRI exam
* Known Hypersensitivity to the active substance or to any of the excipients in Regadenoson or GE-267
* Any contraindication to aminophylline or theophylline: hypotension, unstable cardiac arrhythmias and acute coronary symptoms
* Unstable angina that has not been stabilized with medical therapy
* Severe hypotension
* Decompensated states of heart failure
* Severe Arrhythmias
* Contraindication to the cardiac MRI examination (e.g. inability to hold breath; severe claustrophobia, metallic devices such as pace makers)
* Second or third degree atrioventricular (AV) block or sinus node dysfunction, unless these patients have a functioning artificial pacemaker
* Known pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from which the groups or cohorts will be selected are adults with known or suspected coronary artery disease located in Brandenburg or Mecklenburg-Western Pomerania. Either they already participated in the HerzCheck-Trial (NCT05122793) or they are referred from local cardiologists.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detect mycocardial perfusion defect | at baseline
  Presence of a myocardial perfusion defect indicating significant CAD per participant on GE-267-enhanced cMRI using Regadenoson (detected by visual assessment and/or quantitative perfusion)
Evaluate the image quality of GE-267 | at baseline
  Signal intensity of GE-267 meglumine during perfusion cardiovascular magnetic resonance (detected by quantitative assessment by a score system by two experienced readers and/or image quality assessment by Philips software (SNR/CNR))

SECONDARY OUTCOMES:
Recommendation of the patient to further procedure | 6-8 months
  Recommendation of the patient to further procedure into following classes:
  I) Unremarkable stress-cMRI -> Follow Up of the patient by phone call II) Unremarkable stress-cMRI, but pathologic abnormal MRI -> recommendation for further diagnostic -> Follow Up of the patient by phone call III) Positive stress-cMRI -> recommendation for invasive diagnostic -> Follow Up of the patient by phone call
Comparison of stress-cMRI result and result of invasive diagnostic | 6-8 months
  Comparison of Group with positive stress-cMRI (and recommendation for invasive diagnostic as well as Follow Up of the patient by phone call 6-8 months after MRI): Stress-cMRI result and result of invasive diagnostic
Total examination time | within 2 hours after baseline
  Total examination time including time patient in, examination, patient out time
Adverse Effects | within 2 hours after baseline
  Number of Patients with Any (One or More) Regadenoson and/or GE-267-related Adverse-effect

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Kelle, Prof. Dr., Principal Investigator — Deutsches Herzzentrum der Charité
Locations (1):
- Deutsches Herzzentrum der Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nagel E, Klein C, Paetsch I, Hettwer S, Schnackenburg B, Wegscheider K, Fleck E. Magnetic resonance perfusion measurements for the noninvasive detection of coronary artery disease. Circulation. 2003 Jul 29;108(4):432-7. doi: 10.1161/01.CIR.0000080915.35024.A9. Epub 2003 Jul 14. PMID 12860910
- [Background] Hundley WG, Hamilton CA, Thomas MS, Herrington DM, Salido TB, Kitzman DW, Little WC, Link KM. Utility of fast cine magnetic resonance imaging and display for the detection of myocardial ischemia in patients not well suited for second harmonic stress echocardiography. Circulation. 1999 Oct 19;100(16):1697-702. doi: 10.1161/01.cir.100.16.1697. PMID 10525488
- [Background] Kelle S, Roes SD, Klein C, Kokocinski T, de Roos A, Fleck E, Bax JJ, Nagel E. Prognostic value of myocardial infarct size and contractile reserve using magnetic resonance imaging. J Am Coll Cardiol. 2009 Nov 3;54(19):1770-7. doi: 10.1016/j.jacc.2009.07.027. PMID 19874990
- [Background] Tschope C, Ammirati E, Bozkurt B, Caforio ALP, Cooper LT, Felix SB, Hare JM, Heidecker B, Heymans S, Hubner N, Kelle S, Klingel K, Maatz H, Parwani AS, Spillmann F, Starling RC, Tsutsui H, Seferovic P, Van Linthout S. Myocarditis and inflammatory cardiomyopathy: current evidence and future directions. Nat Rev Cardiol. 2021 Mar;18(3):169-193. doi: 10.1038/s41569-020-00435-x. Epub 2020 Oct 12. PMID 33046850
- [Background] Weiss KJ, Nasser SB, Bigvava T, Doltra A, Schnackenburg B, Berger A, Anker MS, Stehning C, Doeblin P, Abdelmeguid M, Talat M, Gebker R, E-Naggar W, Pieske B, Kelle S. Long-term prognostic value of vasodilator stress cardiac magnetic resonance in patients with atrial fibrillation. ESC Heart Fail. 2022 Feb;9(1):110-121. doi: 10.1002/ehf2.13736. Epub 2021 Dec 6. PMID 34866358
- [Background] Sengupta PP, Kramer CM, Narula J, Dilsizian V. The Potential of Clinical Phenotyping of Heart Failure With Imaging Biomarkers for Guiding Therapies: A Focused Update. JACC Cardiovasc Imaging. 2017 Sep;10(9):1056-1071. doi: 10.1016/j.jcmg.2017.07.001. PMID 28882290
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Background] Kramer CM, Barkhausen J, Bucciarelli-Ducci C, Flamm SD, Kim RJ, Nagel E. Standardized cardiovascular magnetic resonance imaging (CMR) protocols: 2020 update. J Cardiovasc Magn Reson. 2020 Feb 24;22(1):17. doi: 10.1186/s12968-020-00607-1. PMID 32089132
- [Background] Pavon AG, Porretta AP, Arangalage D, Domenichini G, Rutz T, Hugelshofer S, Pruvot E, Monney P, Pascale P, Schwitter J. Feasibility of adenosine stress cardiovascular magnetic resonance perfusion imaging in patients with MR-conditional transvenous permanent pacemakers and defibrillators. J Cardiovasc Magn Reson. 2022 Jan 13;24(1):9. doi: 10.1186/s12968-021-00842-0. PMID 35022037
- [Background] Doltra A, Skorin A, Hamdan A, Schnackenburg B, Gebker R, Klein C, Nagel E, Fleck E, Kelle S. Comparison of acquisition time and dose for late gadolinium enhancement imaging at 3.0 T in patients with chronic myocardial infarction using Gd-BOPTA. Eur Radiol. 2014 Sep;24(9):2192-200. doi: 10.1007/s00330-014-3213-y. Epub 2014 May 15. PMID 24828537